CLINICAL TRIAL: NCT01674634
Title: A Phase 3b Open-label, Historically-controlled Study to Assess the Safety and Efficacy of Two Concurrent Injections of AA4500 in Adult Subjects With Multiple Dupuytren's Contractures With Palpable Cords
Brief Title: Safety and Efficacy of Two Concurrent Injections of AA4500 in Adult Subjects With Multiple Dupuytren's Contractures
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Endo Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AUX-CC-867
Record Dates: First submitted 2012-08-27; First posted 2012-08-29 (Estimated); Results first posted 2015-02-20 (Estimated); Last update posted 2017-10-05 (Actual); Status verified 2017-09

CONDITIONS: Dupuytren's Contracture
Keywords: XIAFLEX; XIAPEX; Dupuytren's disease; contracture
MeSH Terms: conditions — Dupuytren Contracture; Contracture | interventions — Microbial Collagenase; xiapex

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- XIAFLEX / XIAPEX (Experimental): AA4500 (collagenase clostridium histolyticum)
  Interventions: Biological: XIAFLEX / XIAPEX

INTERVENTIONS:
Biological: XIAFLEX / XIAPEX — injection (0.58 mg after reconstitution with sterile diluent [0.3 mg/mL calcium chloride dihydrate in 0.9% sodium chloride])
  Other Names: AA4500 (collagenase clostridium histolyticum)

SUMMARY:
The primary objective of this study is to assess the safety of two concurrent injections of AA4500 into the same hand in subjects with multiple Dupuytren's contractures with palpable cords followed 24 to 72 hours later by a finger extension procedure and compare the rate of occurrence of targeted serious adverse events (tendon rupture/ligament injury and anaphylaxis) to historical rates of the same in clinical studies and post-marketing commercial use.

The secondary objective is to evaluate the efficacy of two concurrent injections of AA4500.

DETAILED DESCRIPTION:
Methodology/Study Design: After all pre-injection procedures are completed on Day 1, eligible men and women will receive two concurrent injections AA4500 (AA4500/AA4500) into cord(s) affecting MP and/or PIP joints on the same or different fingers in the selected hand. A finger extension procedure to facilitate cord disruption will be performed (after administration of local anesthesia, if needed) 24 to 72 hours after injection in those subjects who do not have spontaneous disruption of their cord(s).

Follow up visits for the evaluation of safety and efficacy will be required for all subjects 24 to 72 hours after injection, and on Days 15, 31, and 61.

Upon completion of the day 61 follow-up visit (end of study visit), subjects who require additional treatment in the treated hand may receive up to three additional injections of AA4500 according to the XIAFLEX package insert. Subjects may receive up to a total of five injections and individual cords may receive up to a total of three injections. Subjects who require additional treatment will be followed for safety.

ELIGIBILITY:
Inclusion Criteria:

1. Provide a signed and dated informed consent
2. Be a man or woman ≥ 18 years of age
3. Have a diagnosis of Dupuytren's disease and have at least 2 fixed-flexion contractures on the same hand that are ≥ 20º in PIP and/or MP joints in fingers, other than the thumbs, which are caused by palpable cord(s) suitable for treatment
4. Have a positive "table top test" defined as the inability to simultaneously place the affected finger(s) and palm flat against a table top
5. Have a negative urine pregnancy test at screening and before injection of study drug and be using a highly effective (ie, < 1% failure rate) contraception method as judged by the investigator (eg, abstinence, intrauterine device [IUD], hormonal [estrogen/progestin] contraceptives, or barrier control) for at least one menstrual cycle prior to study enrollment and for the duration of the study or be surgically sterile (if female of childbearing potential); or be a postmenopausal female (no menses for at least 1 year or hysterectomy).
6. Be able to comply with the study visit schedule as specified in the protocol

Exclusion Criteria:

A subject will be excluded from study participation if he/she:

1. Received surgery (fasciectomy or surgical fasciotomy) and/or needle aponeurotomy/fasciotomy on the selected joints to be treated within 6 months before administration of study drug
2. Has a chronic muscular, neurological, or neuromuscular disorder that affects the hands
3. Has a known systemic allergy to collagenase or any other excipient of AA4500
4. Has received any collagenase treatments (eg, Santyl® ointment and/or XIAFLEX®/XIAPEX®) within 30 days before injection of study drug in the hand selected for treatment
5. Is currently receiving or plans to receive anticoagulant medication or has received anticoagulant medication (except for ≤ 150 mg aspirin daily) within 7 days before injection of study drug
6. Has a known recent history of stroke, bleeding, or other medical condition, which in the investigator's opinion would make the subject unsuitable for enrollment in the study
7. Received an investigational drug within 30 days before injection of study drug
8. Is pregnant or intends on becoming pregnant during the study or is breastfeeding a child
9. Has any clinically significant medical history or condition(s), including conditions that affect the hands, that would, in the opinion of the investigator, substantially increase the risk associated with the subject's participation in the protocol or compromise the scientific objectives of the study
10. Has jewelry on the hand to be treated that cannot be removed

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 715 (Actual)
Dates: Start 2012-09; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Veronica Urdaneta, MD, MPPH, Study Director — Endo Pharmaceuticals
Locations (25):
- United States (25):
  - HOPE Research Institute, Phoenix, Arizona
  - Tucson Orthopaedic Institute, Tucson, Arizona
  - CORE Orthopaedic Medical Center, Encinitas, California
  - Torrey Pines Medical Group, La Jolla, California
  - Brigid Freyne, MD, Inc., Murrieta, California
  - The Hand and Upper Extremity Center, Atlanta, Georgia
  - Rockford Orthopedic Associates, Rockford, Illinois
  - The Indiana Hand to Shoulder Center, Indianapolis, Indiana
  - University of Kansas Medical Center, Kansas City, Kansas
  - Christine M. Kleinert Institute for Hand and Microsurgery, Inc., Louisville, Kentucky
  - Lake Cumberland Rheumatology, Somerset, Kentucky
  - TRIA Orthopedic Center, Minneapolis, Minnesota
  - Missoula Bone and Joint, Missoula, Montana
  - Nevada Orthopedic and Spine Center, Las Vegas, Nevada
  - Central Jersey Hand Surgery, Eatontown, New Jersey
  - Hospital for Special Surgery, New York, New York
  - SUNY Stony Brook, Setauket, New York
  - UNC School of Medicine, Chapel Hill, North Carolina
  - OrthoCarolina Research Institute, Inc., Charlotte, North Carolina
  - Health Research Institute, Oklahoma City, Oklahoma
  - The Center for Neurosurgical and Orthopedic Care and Research, Bend, Oregon
  - Hand Microsurgery & Reconstructive Orthopaedics, Erie, Pennsylvania
  - Alpha Clinical Research, LLC, Clarksville, Tennessee
  - Accurate Clinical Research, Inc., Houston, Texas
  - The Arthritis Clinic of Northern Virginia, PA, Arlington, Virginia

RESULTS

PARTICIPANT FLOW:
Groups:
- XIAFLEX/XIAPEX: AA4500 (collagenase clostridium histolyticum): 2 concurrent 0.58 mg injections (1 injection per joint) in the same hand
Period: Overall Study
Arm/Group | XIAFLEX/XIAPEX
Started | 715
Completed | 709
Not Completed | 6
Not completed — Withdrawal by Subject | 3
Not completed — Lost to Follow-up | 3

BASELINE CHARACTERISTICS:
Arm/Group | XIAFLEX/XIAPEX
Number analyzed (Participants) | 715
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 348
  >=65 years | 367
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.0 (9.26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 99
  Male | 616
Region of Enrollment [Number; unit: participants]
  United States | 278
  Australia | 196
  New Zealand | 70
  Denmark | 87
  Sweden | 50
  United Kingdom | 34

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Total Fixed Flexion
Description: Percent change from baseline in total fixed flexion = 100 * (baseline total FFC - day 31 total FFC)/baseline total FFC, where total fixed flexion is defined as the sum of the fixed flexion contracture (FCC) of the 2 joints receiving treatment. Positive percent change from baseline indicates improvement.
Time Frame: Baseline, Day 31
Population: Efficacy analysis was based on the modified intent-to-treat (mITT) population; all enrolled subjects who received both AA4500 injections and had a post-injection efficacy measure. Ten subjects were granted special re-enrollment and had an additional joint pair treated on contralateral hand. Assessment is based on simultaneously treated joint pairs.
Measure: Mean (Standard Deviation); unit: percentage of contracture change
Units Other Than Participants: Treated Joint Pairs
Arm/Group | XIAFLEX/XIAPEX
Number analyzed (Participants) | 714
Number analyzed (Treated Joint Pairs) | 724
percentage of contracture change | 74.41 (24.83)

2. Primary Outcome: Change From Baseline in Total Range of Motion
Description: The total range of motion (ROM) is the sum of the range of motion measurements of the 2 treated joints. ROM is defined as difference between full flexion angle and full extension expressed in degrees. A positive change from baseline indicates increased (improved) ROM.
Time Frame: Baseline, Day 31
Population: Efficacy analysis was based on the mITT population; all enrolled subjects who received both AA4500 injections and had a post-injection efficacy measure. Ten subjects were granted special re-enrollment and had an additional joint pair treated on the contralateral hand. Assessment is based on simultaneously treated joint pairs.
Measure: Mean (95% Confidence Interval); unit: degrees
Units Other Than Participants: treated joint pairs
Arm/Group | XIAFLEX/XIAPEX
Number analyzed (Participants) | 714
Number analyzed (treated joint pairs) | 724
degrees | 66.6 [64.3 to 68.9]

3. Secondary Outcome: Clinical Success
Description: Clinical success is defined as reduction of FFC of a treated joint to within 0-5 degrees of normal within 30 days of injection
Time Frame: Within 30 days
Population: Efficacy analysis was based on the mITT population; all enrolled subjects who received both AA4500 injections and had a post-injection efficacy measure. Ten subjects were granted special re-enrollment and had an additional joint pair treated on the contralateral hand. This assessment is based on individual treated joints by joint type.
Measure: Number; unit: Joints
Units Other Than Participants: Treated Joints
Groups:
- XIAFLEX/XIAPEX MP Joint: AA4500 (collagenase clostridium histolyticum); 0.58 mg injection in the metacarpophalangeal (MP) joint cord
- XIAFLEX/XIAPEX PIP Joint: AA4500 (collagenase clostridium histolyticum); 0.58 mg injection in the proximal interphalangeal (PIP) joint cord
Arm/Group | XIAFLEX/XIAPEX MP Joint | XIAFLEX/XIAPEX PIP Joint
Number analyzed (Participants) | 714 | 714
Number analyzed (Treated Joints) | 896 | 552
Joints
  No | 317 | 394
  Yes | 579 | 158

4. Secondary Outcome: Clinical Improvement
Description: Clinical improvement is defined as a reduction of FFC by 50% or greater of the baseline value within 30 days of injection
Time Frame: Within 30 days
Population: as for outcome 3
Measure: Number; unit: Joints
Units Other Than Participants: Treated Joints
Groups:
- XIAFLEX/XIAPEX MP Joint: AA4500 (collagenase clostridium histolyticum); 0.58 mg injection in the MP joint cord
- XIAFLEX/XIAPEX PIP Joint: AA4500 (collagenase clostridium histolyticum); 0.58 mg injection in the PIP joint cord
Arm/Group | XIAFLEX/XIAPEX MP Joint | XIAFLEX/XIAPEX PIP Joint
Number analyzed (Participants) | 714 | 714
Number analyzed (Treated Joints) | 896 | 552
Joints
  No | 96 | 157
  Yes | 800 | 395

5. Secondary Outcome: Subject Assessment of Satisfaction With Treatment at Day 31
Description: Subject's were asked to rate satisfaction with treatment at the day 31 follow-up visit
Time Frame: Day 31
Population: as for outcome 2
Measure: Number; unit: Joint Pairs
Units Other Than Participants: Treated Joint Pairs
Arm/Group | XIAFLEX/XIAPEX
Number analyzed (Participants) | 714
Number analyzed (Treated Joint Pairs) | 724
Joint Pairs
  Very satisfied | 461
  Quite satisfied | 198
  Neither satisfied nor dissatisfied | 38
  Quite dissatisfied | 9
  Very dissatisfied | 6
  Not done | 12

6. Secondary Outcome: Subject Assessment of Satisfaction With Treatment at Day 61
Description: Subject's were asked to rate satisfaction with treatment at the day 61 follow-up visit
Time Frame: Day 61
Population: as for outcome 2
Measure: Number; unit: Joint Pairs
Units Other Than Participants: Treated Joint Pairs
Arm/Group | XIAFLEX/XIAPEX
Number analyzed (Participants) | 714
Number analyzed (Treated Joint Pairs) | 724
Joint Pairs
  Very satisfied | 496
  Quite satisfied | 167
  Neither satisfied nor dissatisfied | 38
  Quite dissatisfied | 11
  Very dissatisfied | 8
  Not done | 4

7. Secondary Outcome: Investigator Assessment of Improvement With Treatment at Day 31
Description: Investigator's determined the degree of improvement in the severity of the subject's treated finger(s) compared with screening at the day 31 follow-up visit.
Time Frame: Day 31
Population: as for outcome 2
Measure: Number; unit: Joint Pairs
Units Other Than Participants: Treated Joint Pairs
Arm/Group | XIAFLEX/XIAPEX
Number analyzed (Participants) | 714
Number analyzed (Treated Joint Pairs) | 724
Joint Pairs
  Very much improved | 375
  Much improved | 271
  Minimally improved | 51
  No change | 4
  Minimally worse | 3
  Much worse | 0
  Very much worse | 0
  Not done | 20

8. Secondary Outcome: Investigator Assessment of Improvement With Treatment at Day 61
Description: Investigator's determined the degree of improvement in the severity of the subject's treated finger(s) compared with screening at the day 61 follow-up visit.
Time Frame: Day 61
Population: as for outcome 2
Measure: Number; unit: Joint Pairs
Units Other Than Participants: Treated Joint Pairs
Arm/Group | XIAFLEX/XIAPEX
Number analyzed (Participants) | 714
Number analyzed (Treated Joint Pairs) | 724
Joint Pairs
  Very much improved | 382
  Much improved | 263
  Minimally improved | 62
  No change | 7
  Minimally worse | 2
  Much worse | 0
  Very much worse | 0
  Not done | 8

9. Secondary Outcome: Change From Baseline for Unité Rhumatologique Des Affections de la Main Scale at Day 31
Description: The Unité Rhumatologique des Affections de la Main (URAM) scale is a patient-reported functional 9-item scale (total score 0-45) developed and validated to assess functional outcome of patients suffering from Dupuytren's disease with higher scores indicating greater difficulty using the hand.The estimated clinically important change of the URAM scale is 2.9 points. A decrease in total URAM score indicates improvement in hand function.
Time Frame: Baseline, Day 31
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Treated Joint Pairs
Arm/Group | XIAFLEX/XIAPEX
Number analyzed (Participants) | 714
Number analyzed (Treated Joint Pairs) | 724
units on a scale | -11.3 (9.19)

10. Secondary Outcome: Change From Baseline for Unité Rhumatologique Des Affections de la Main Scale at Day 61
Description: The URAM scale is a patient-reported functional 9-item scale (total score 0-45) developed and validated to assess functional outcome of patients suffering from Dupuytren's disease with higher scores indicating greater difficulty using the hand.The estimated clinically important change of the URAM scale is 2.9 points. A decrease in total URAM score indicates improvement in hand function.
Time Frame: Baseline, Day 61
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Treated Joint Pairs
Arm/Group | XIAFLEX/XIAPEX
Number analyzed (Participants) | 714
Number analyzed (Treated Joint Pairs) | 724
units on a scale | -12.3 (9.75)

ADVERSE EVENTS:
Arm/Group | XIAFLEX/XIAPEX
Serious Adverse Events (participants affected / at risk) | 15/715
Other Adverse Events (participants affected / at risk) | 680/715
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | XIAFLEX/XIAPEX (N=715)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 1 (1)
Feeding tube complication (Injury, poisoning and procedural complications) | 1 (1) — PEG feeding tube obstruction
Arteriosclerosis (Vascular disorders) | 1 (1)
Myelopathy (Nervous system disorders) | 1 (1)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) — Bleeding left hand post procedure
Lymphangitis (Infections and infestations) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1)
Malaise (General disorders) | 1 (1)
oedema peripheral (General disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Anal abscess (Infections and infestations) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) — Left lower leg
Tendon rupture (Injury, poisoning and procedural complications) | 1 (1) — Upgraded to an SAE by the sponsor
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | XIAFLEX/XIAPEX (N=715)
Oedema peripheral (General disorders) | 552 (626)
Contusion (Injury, poisoning and procedural complications) | 420 (513)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 361 (431)
Laceration (Injury, poisoning and procedural complications) | 184 (192)
Pruritus (Skin and subcutaneous tissue disorders) | 107 (121)
Injection site pain (General disorders) | 102 (109)
Lymphadenopathy (Blood and lymphatic system disorders) | 92 (102)
Blood blister (Skin and subcutaneous tissue disorders) | 89 (98)
Injection site haematoma (General disorders) | 60 (61)
Axillary pain (General disorders) | 51 (53)
injection site haemorrhage (General disorders) | 45 (45) — injection site ecchymosis
Injection site swelling (General disorders) | 42 (42)
Ecchymosis (Skin and subcutaneous tissue disorders) | 37 (39)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other